CLINICAL TRIAL: NCT04173065
Title: VK2809 A Phase 2B, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to Assess the Efficacy, Safety, and Tolerability of VK2809 Administered for 52 Weeks Followed by a 4-Week Off-Drug Phase in Subjects With Biopsy Proven Non-Alcoholic Steatohepatitis With Fibrosis
Brief Title: A Study to Assess the Efficacy and Safety of VK2809 for 52 Weeks in Subjects With Biopsy Proven NASH
Acronym: VOYAGE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Viking Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VK2809-202
Record Dates: First submitted 2019-11-20; First posted 2019-11-21 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: NASH - Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — 2-((3,5-dimethyl-4-(4'-hydroxy-3'-isopropylbenzyl)phenoxy)methyl)-4-(3-chlorophenyl)-2-oxido(1,3,2)dioxaphosphonane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebos
- 1.0 mg (Experimental)
  Interventions: Drug: VK2809
- 2.5mg (Experimental)
  Interventions: Drug: VK2809
- 5.0 mg (Experimental)
  Interventions: Drug: VK2809
- 10 mg (Experimental)
  Interventions: Drug: VK2809

INTERVENTIONS:
Drug: VK2809 — Capsule
  Arms: 1.0 mg; 10 mg; 2.5mg; 5.0 mg
Drug: Placebos — Capsule
  Arms: Placebo

SUMMARY:
The study includes 52 weeks, double-blind treatment period. Clinic visits will occur at Randomization and every four weeks from Week 4 through Week 52 and through End of Study period. The study includes a post-dosing study visit that will occur 4 weeks after the last dose of study drug. This visit represents the End-of-Study Visit (Week 56 Visit). Three hundred thirty-seven subjects will be enrolled into five treatment arms and there will be an equal distribution of males and females in each treatment arm. Subjects will be stratified by gender, fibrosis stage, and diabetes status.

ELIGIBILITY:
Inclusion Criteria:

1. Provide a personally signed and dated informed consent document indicating that the subject (or a legally acceptable representative) has been informed of all pertinent aspects of the study and is willing and able to participate;
2. Have a histologically-confirmed diagnosis of NASH on a liver biopsy performed during screening or within 6 months before screening; for this study, confirmation requires:

   1. NASH Clinical Research Network (CRN) fibrosis stage 1 to stage 3 and
   2. NASH activity score (NAS) of ≥4 with at least a score of 1 in each of the following NAS components: ballooning degeneration (score = 0-2), lobular inflammation (score = 0-3) and steatosis (score = 0-3); (c) F1 subjects must have at least one of these risk factors: type 2 diabetes, body mass index of ≥ 30 mg/ m2, and/ or alanine aminotransferase > 1.5 x ULN
3. Have a screening MRI-PDFF with ≥ 8% liver fat fraction;
4. Male and females be 18 to 75 years of age, inclusive, at screening;

Exclusion Criteria:

1. Are unwilling to undergo the required liver biopsy procedures or have any condition that would prevent obtaining a liver biopsy as part of this clinical protocol
2. Have evidence of current or history of excessive alcohol consumption of more than 20 g per day for women and 30 g per day for men, on average, within 6 months before the qualifying liver biopsy and up to randomization, or are unable to provide a reliable estimate of alcohol consumption during this period;
3. Treatment with medications for the purpose of weight loss within 6 months prior to qualifying liver biopsy, unless approved after consultation with the medical monitor. These include drugs approved for weight loss (e.g. orlistat, bupropion/naltrexone, phentermine-topiramate, phentermine, lorcaserin), as well as drugs used off-label, herbal preparations and dietary supplements marketed for control of body weight or appetite;
4. TSH outside central laboratory reference range;
5. Free T4 outside central laboratory reference range;
6. Cardiac troponin I (cTnI) and creatine kinase MB isoenzyme (CK-MB) > Upper Limit of Normal (ULN) at screening;
7. Serum albumin < 3.5 g/dL;
8. International normalized ratio (INR) > 1.3;
9. Total bilirubin > 1.2 X ULN (except in presence of Gilbert synd
10. Strong or moderate inhibitors or inducers of CYP3A4 are prohibited during the study period
11. Drugs that may affect liver fat content or are associated with nonalcoholic fatty liver disease (NAFLD) are prohibited during the 3 month period prior to the baseline liver biopsy and up to the end of treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2024-01-26 (Actual)

PRIMARY OUTCOMES:
Liver Fat | 12 weeks
  Relative change in liver fat content (assessed by MRI-PDFF) from baseline to Week 12 in subjects treated with VK2809 compared to the change in subjects treated with placebo.

SECONDARY OUTCOMES:
NASH CRN fibrosis score | 52 weeks
  Proportion of subjects with resolution of steatohepatitis on overall histopathological reading and no worsening of liver fibrosis on NASH CRN fibrosis score.

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Mancini, MA, MBA, Study Director — Viking Therapeutics, Inc.
Locations (79):
- United States (68):
  - Viking Clinical Site 105, Madison, Alabama
  - Viking Clinical Site 216, Glendale, Arizona
  - Viking Clinical Site 159, Tucson, Arizona
  - Viking Clinical Site 214, North Little Rock, Arkansas
  - Viking Clinical Site 161, Fresno, California
  - Viking Clinical Site 208, Fresno, California
  - Viking Clinical Site 302, La Jolla, California
  - Viking Clinical Site 134, Montclair, California
  - Viking Clinical Site 205, Panorama City, California
  - Viking Clinical Site 125, Pasadena, California
  - Viking Clinical Site 110, Rialto, California
  - Viking Clinical Site 117, Sacramento, California
  - Viking Clinical Site 121, San Diego, California
  - Viking Clinical Site 103, San Francisco, California
  - Viking Clinical Site 156, New Haven, Connecticut
  - Viking Clinical Site 226, Bradenton, Florida
  - Viking Clinical Site 150, Lakewood Rch, Florida
  - Viking Clinical Site 106, Miami, Florida
  - Viking Clinical Site 301, Miami, Florida
  - Viking Clinical Site 310, Miami, Florida
  - Viking Clinical Site 221, Miami Lakes, Florida
  - Viking Clinical Site 131, Pensacola, Florida
  - Viking Clinical Site 215, Port Orange, Florida
  - Viking Clinical Site 218, Sarasota, Florida
  - Viking Clinical Site 144, Atlanta, Georgia
  - Viking Clinical Site 111, Marietta, Georgia
  - Viking Clinical Site 120, Indianapolis, Indiana
  - Viking Clinical Site 130, South Bend, Indiana
  - Viking Clinical Site 211, West Des Moines, Iowa
  - Viking Clinical Site 145, Topeka, Kansas
  - Viking Clinical Site 146, Marrero, Louisiana
  - Viking Clinical Site 307, New Orleans, Louisiana
  - Viking Clinical Site 166, West Monroe, Louisiana
  - Viking Clinical Site 109, Baltimore, Maryland
  - Viking Clinical Site 107, Greenbelt, Maryland
  - Viking Clinical Site 147, Boston, Massachusetts
  - Viking Clinical Site 158, Ann Arbor, Michigan
  - Viking Clinical Site 133, Detroit, Michigan
  - Viking Clinical Site 213, Jackson, Mississippi
  - Viking Clinical Site 112, Kansas City, Missouri
  - Viking Clinical Site 217, Kansas City, Missouri
  - Viking Clinical Site 160, Las Vegas, Nevada
  - Viking Clinical Site 223, Reno, Nevada
  - Viking Clinical Site 152, New York, New York
  - Viking Clinical Site 128, Rochester, New York
  - Viking Clinical Site 314, Chapel Hill, North Carolina
  - Viking Clinical Site 126, Concord, North Carolina
  - Viking Clinical Site 116, Durham, North Carolina
  - Viking Clinical Site 153, Morehead City, North Carolina
  - Viking Clinical Site 137, Cincinnati, Ohio
  - Viking Clinical Site 148, Philadelphia, Pennsylvania
  - Viking Clinical Site 311, Pittsburgh, Pennsylvania
  - Viking Clinical Site 127, Greenville, South Carolina
  - Viking Clinical Site 227, Clarksville, Tennessee
  - Viking Clinical Site 118, Hermitage, Tennessee
  - Viking Clinical Site 115, Arlington, Texas
  - Viking Clinical Site 113, Dallas, Texas
  - Viking Clinical Site 220, Edinburg, Texas
  - Viking Clinical Site 142, Houston, Texas
  - Viking Clinical Site 102, San Antonio, Texas
  - Viking Clinical Site 101, San Antonio, Texas
  - Viking Clinical Site 143, San Antonio, Texas
  - Viking Clinical Site 201, San Antonio, Texas
  - Viking Clinical Site 224, Ogden, Utah
  - Viking Clinical Site 304, Newport News, Virginia
  - Viking Clinical Site 209, Richmond, Virginia
  - Viking Clinical Site 312, Richmond, Virginia
  - Viking Clinical Site 317, Seattle, Washington
- Belgium (2):
  - Viking Clinical Site 503, Brussels, VBR
  - Viking Clinical Site 502, Brussels
- France (5):
  - Viking Clinical Site 611, Amiens
  - Viking Clinical Site 612, Créteil
  - Viking Clinical Site 610, Grenoble
  - Viking Clinical Site 607, Paris
  - Viking Clinical Site 603, Paris
- Mexico (3):
  - Viking Clinical Site 401, Acapulco de Juárez, Guerrero
  - Viking Clinical Site 422, Monterrey, Nuevo León
  - Viking Clinical Site 421, Mexico City
- Viking Clinical Site 219, San Juan, Puerto Rico